CLINICAL TRIAL: NCT07251647
Title: Adaptation of the Mini-Mental State Examination (MMSE) for the Reunion Island Population
Acronym: MMSE-RUN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025/CHU/10
Record Dates: First submitted 2025-10-02; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Alzheimer s Disease; Vascular Cognitive Impairment
Keywords: Neurocognitive disorder; cognitive test; screening; Reunion Island
MeSH Terms: conditions — Neurocognitive Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (Healthy indivuduals) (Other): MMSE-RUN and MMSE GRECO questionnaires
  Interventions: Diagnostic Test: MMSE-RUN and MMSE GRECO
- Case Arm (Patients with Alzheimer's disease or vascular cognitive impairment) (Other): MMSE-RUN and MMSE GRECO questionnaires
  Interventions: Diagnostic Test: MMSE-RUN and MMSE GRECO

INTERVENTIONS:
Diagnostic Test: MMSE-RUN and MMSE GRECO — Each participant (control and Case) will complete MMSE-RUN and MMSE-GRECO.

SUMMARY:
The Mini-Mental State Examination (MMSE) is the most widely used cognitive screening and monitoring test for neurocognitive disorders in current clinical practice. Its French version was published in 1998 by the GRECO group (MMSE-GRECO). However, some items of this French version are not adapted to local Reunionese particularities.

The main objective is to propose and validate the psychometric properties of an adapted version of the MMSE, to the Reunionese culture (MMSE-RUN) in a healthy population and in a sick population (Alzheimer's Disease and Vascular Cognitive Disorder), and to compare its performance with the MMSE-GRECO.

DETAILED DESCRIPTION:
The MMSE score was described in 1975 by an American psychiatrist. Due to its good psychometric properties and its quick and simple administration, it has become the most widely known and used screening and monitoring test for neurocognitive disorders. The MMSE have been translated and adapted for use in many languages and cultures worldwide. Its brevity, ease of use, and established psychometric properties have contributed to its widespread adoption in clinical practice and research settings for detecting cognitive impairment and monitoring cognitive changes over time.

It has been adapted into French (MMSE-GRECO), as well as to other cultures in Europe, Asia, and Africa. In the French overseas territories, a Polynesian and Caribbean version have been published.

In Reunion Island, no adapted version has been published yet. Nevertheless, an early identification of cognitive disorders with adapted screening tools is essential because three risk factors for cognitive vulnerability converge: (1) an aging population (increasing the risk of developing Alzheimer's disease) with (2) a lower level of education (decreasing cognitive resilience), and (3) a higher frequency of cardiovascular risk factors (hypertension, diabetes, dyslipidemia), increasing the frequency of vascular cognitive disorders.

The objective of this study is to propose an adapted version of the test for the Reunion Island population (MMSE-RUN) and to validate its psychometric properties within a cohort of healthy subjects and patients (Alzheimer's disease and/or vascular cognitive disorder).

ELIGIBILITY:
Inclusion criteria:

* For the healthy population : aged 60 to 89 years, residing in Reunion for more than 5 years, able to understand the test instructions, available for a one-hour interview, affiliated with a social security scheme, with informed consent.
* For the sick population : aged 60 to 89 years, residing in Reunion for more than 5 years, presenting probable or possible Alzheimer's disease and/or probable vascular cognitive disorder, able to understand the test instructions, available for a one-hour interview, affiliated with a social security scheme, with informed consent.

Exclusion criteria:

* For the healthy populationhistory of neurological pathology, neurodegenerative pathology with cognitive expression, refusing to participate in the study, under legal protection.
* For the sick population: acute unresolved medical decompensation or acute psychic decompensation, refusing to participate in the study, under legal protection.

Ages: 60 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Internal consistency - Cronbach's alpha | Day 1
  Internal consistency measures the extent to which the items in the test measure the same dimension or concept, in this case overall cognitive efficiency.
  Internal consistency is commonly measured by Cronbach's alpha, which ranges from 0 (low) to 1 (high). A high coefficient indicates that the test items are similar in content, i.e. homogeneous. A Cronbach's alpha greater than 0.7 is acceptable.
Construct validity - Exploratory Factor Analysis | Day 1
  Construct validity allows us to visualise the construction of the test and the concept measured by the instrument in healthy population. The existence of seven independent factors must be demonstrated by Exploratory Factor Analysis: temporal orientation, spatial orientation, learning three words, mental arithmetic, recall, language and constructive praxis.
Criterion validity - t test | Day 1
  Criterion validity consists of verifying an instrument's ability to distinguish between individuals; ie, it is the test's ability to clearly identify a deficit in overall cognitive efficiency in a population affected by a pathology, compared to a cognitively healthy population.
  The validity of this criterion will be assessed using a Student's t-test comparing the MMSE-RUN scores obtained by the healthy subjects group and the pathological subjects group.

CONTACTS AND LOCATIONS:
Locations (7):
- Reunion (7):
  - CHU de La Réunion - site Nord - Geriatric department, Saint-Denis
  - CHU de La Réunion - site Nord - Neurology department, Saint-Denis
  - Centre Hospitalier Ouest Réunion (CHOR), Saint-Paul
  - CHU de La Réunion - site Sud - Geriatric department, Saint-Pierre
  - CHU de La Réunion - site Sud - Neurology department, Saint-Pierre
  - CHU de La Réunion, Saint-Pierre
  - Functional Rehabilitation Center, Sainte-Clotilde

IPD SHARING:
Plan to Share IPD: No